CLINICAL TRIAL: NCT03613896
Title: Accuracy of 3D Printed Maxillary Complete Dentures Compared With Conventional Complete Dentures: Non-Randomized Control Trial
Brief Title: Accuracy of 3D Printed Maxillary Complete Dentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer mohamed mohamed, Principal Investigator, Cairo University
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: hadeer's protocol
Record Dates: First submitted 2018-07-05; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Accuracy of 3d Printed Dentures

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional dentures (Placebo Comparator): a complete denture made through conventional processing technique
  Interventions: Procedure: conventional dentures
- 3D printed dentures (Active Comparator): a complete denture made through 3d printing
  Interventions: Procedure: 3d printed denture

INTERVENTIONS:
Procedure: conventional dentures — conventional dentures
  Arms: conventional dentures
Procedure: 3d printed denture — construction of a 3d printed denture through a recent method instead of conventional heat processing
  Arms: 3D printed dentures

SUMMARY:
Conventional complete dentures have been used for almost a century as a treatment choice for edentulous patients, despite of their inaccuracy & dimensional changes during manufacturing. Recently, new manufacturing techniques like RP/3D printing (rapid prototyping) has progressed in the dental field including prosthodontics, does the 3D printed complete denture show more accuracy than conventional ones?

DETAILED DESCRIPTION:
Conventional complete dentures have been used as a clinically accepted prosthetic treatment for completely edentulous patients for almost a century. [1] One of its advantages is ability to customize teeth arrangement and to check each step of the preceding steps before the delivery stage.

Conventional complete dentures fabrication consist of several steps of recording, transferring, evaluating, and creating artificial substitutes for patient's teeth and gingiva which must be in harmony with patient's mouth and face. All this steps demand high experience, artistic, and skillful operator and technician.

However denture processing results in polymerization shrinkage of the resin (due to flask cooling), and distortion of the denture base (due to stress release after denture base removal from the stone cast), and decreasing the accuracy and denture adaptation. [2] These dimensional changes increase the gap between the denture base and underlying mucosa, resulting in an ill-fitting denture.[3] Denture adaptation and fitting plays a crucial role in complete denture retention (by physical means), stability, and patient comfort. [4]

Also, flask closure must be done under considerable pressure to ensure metal-to-metal contact between the halves of the flask to confine the resin inside the mold with no excess.[5] In addition to the inherent processing shrinkage and/or expansion properties of the acrylic resin.[6] Researchers tried to overcome these disadvantages by changing the technique of polymerization of the resin, by using of microwave energy, dry heat, and visible light.[7] But unfortunately researchers found that, Discrepancies in the base adaptation shown by several techniques are not easily corrected after complete denture processing.[8] Denture base adaptation to the stone cast is usually not satisfactory, especially in the midline section of the central portion of the posterior border.[9] To overcome the previous disadvantages computer aided manufacturing technology was applied to complete dentures. Some advantages of digitally fabricated complete dentures are 1) reduced number of patient visits; 2) superior strength and fit of dentures; 3) omitting multiple error-introducing steps such as impression, waxing, and casting.[10] 4) reduced cost for patient and clinician; 5) easy denture duplication (due to stored digital data); 6) standardization of clinical research on complete dentures and implant-retained overdentures.

To fabricate physical prototype (model) there are two different approaches: subtractive and additive manufacturing.

Subtractive manufacturing is based on milling the denture from a larger blank by a computer numeric controlled (CNC) machine. The input data for this method are principally from an optical or contact probe digitizer, which can only capture the external surface data of the anatomy and not the internal tissue surface of the object.

Although CAD/CAM dentures have many advantages compared to conventional ones, but the CAD/CAM protocol introduces additional steps (like scanning, software modeling, and milling) in the fabrication process that can lead to inaccuracies.[11] Another disadvantage of CAD/CAM is its inability to reproduce fine details by milling .[12] Additive manufacturing is the process that creates objects from 3D model data, in an additive layer by layer manner.[13] The additive systems used in dentistry are stereo-lithography, selective laser sintering or melting, and 3D printing.

The main advantage of additive technology is the ability to create minor details (undercuts, voids, complex internal geometries) in the proposed model. In addition to Incremental vertical object build-up, no material wastage, large objects produced, passive production (i.e., no force application), and ability to print multiple materials at the same time (in case of 3D printing). [15] A clinical study was done to compare the accuracy values of maxillary conventional heat-polymerized trial denture bases with those RR printed ones and the results were as follows: Mean deviation was (-0.0051mm), (SD, 0.19mm).[16]

In the same study authors used ratings from 100-mm VAS in 10 patients and 20 prosthodontists comparing conventional and RP methods and the results were as follows:

Patients comparing overall satisfaction: P=0.59, prosthodontists comparing overall satisfaction: P=0.87 The term selective laser sintering is used to describe the fabrication of a pattern from ceramics or polymers while selective laser melting describes pattern fabrication from metal.[14] The laser beam locally raises the temperature close to the melting point of the metal particle, to avoid complete melting. The platform is slightly immersed in the powder, and powder thickness is controlled by a cylinder rolling on the powder pool. After each new powder layer application, the laser melting process is repeated until the 3D object is completed.

Stereo lithography technology consists of photosensitive resin bath, a model-building platform, and ultraviolet laser for curing. To fabricate the desired model the layers are cured successively, and bonded together from bottom to top. As the first layer is polymerized the model-building platform is brought down inside the bath, and another layer of resin is added and cured. This process continues until the desired model is completed.

In 3D printing system the material is extruded from a nozzle that solidifies as soon as it is deposited on the manufacturing platform. The layer pattern is achieved through horizontal nozzle movement and interrupted material flow. This is followed by vertical movement for the sequential layer deposition.

The captured 3D data of model slice into cross-sections by a certain thickness. Inputting the processing parameters based on the contour information of each layer sheet allows for the automatic generation of the numerical code. Finally, a 3D object consisting of a series of layers is formed by stacking. This technology can receive CAD data directly and create new samples or models quickly without need for molds, cutting tools, or tooling fixtures.

Thanks to this technology, wasting less material, employing less human power, decreasing treatment time at the chair side, decreasing treatment cost, and lowering the rates of contamination, is possible.

In this study, a combination of conventional technique and RP will be used to fabricate complete dentures to overcome the polymerization shrinkage which results from conventional processing.

Explanation for choice of comparators:

Heat processed denture base is the treatment of choice for most of edentulous patients and it is considered as the golden standard and the main comparator for the new techniques. But using Heat Cured Acrylic resin would require many laboratory steps which introduce several errors.[14] Meanwhile, the introduction of rapid prototyping method with high accuracy which eliminates some of the laboratory steps was the reason for choosing it to compare it with the conventional method

ELIGIBILITY:
Inclusion Criteria:

* Cooperative patients with well developed ridges..

Exclusion Criteria:

* Pathological changes of residual ridges.
* Patients with any systemic diseases.
* Patients with xerostomia.
* Patients with flabby and flat ridges.
* Patients with allergy to resins.
* Patient with sever undercuts, or irregular bony exostosis.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy in terms of dimensional changes in denture base | immediately after denture construction
  we will use radio-opaque markers to measure accuracy on software

IPD SHARING:
Plan to Share IPD: Undecided